CLINICAL TRIAL: NCT00628940
Title: PET Imaging of High-grade Glioma Using 18F-fluoromethylcholine: a Tool for the Early Detection of Tumour Recurrence After Combined Radiochemotherapy?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other); Special Research Fund, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008/085
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: High-grade Glioma of the Brain
MeSH Terms: interventions — fluoromethylcholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 18F-fluoromethylcholine
  Interventions: Radiation: PET images with 18F-fluoromethylcholine

INTERVENTIONS:
Radiation: PET images with 18F-fluoromethylcholine — sequential PET images with 18F-fluoromethylcholine

SUMMARY:
The aim of the study is to define preferential sites of tumour recurrence by observing tracer uptake in the tumour in sequential PET images with 18F-fluoromethylcholine (and perfusion MR, see also below). Changes in the intensity of the tracer uptake in the tumour during and after the course of radiotherapy will be correlated with the site of tumour recurrence as will be assessed by conventional MRI. In due time, these results must enable clinicians to change their therapeutic approach of high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* patients with high-grade glioma who will undergo adjuvant radiochemotherapy after surgery

Exclusion Criteria:

* low global performance state
* pregnancy
* lactation period
* presence of pacemaker, vascular clips in the brain ,epidural electrodes, implanted hearing device, set of false theeth attached by means of magnetes, wig attached by means of metal clips

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01-12 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
time to local recurrence after neurosurgery and adjuvant radiochemotherapy | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Goethals, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium